CLINICAL TRIAL: NCT04792463
Title: Frequency and Clinical Phenotype of BAP1 Hereditary Predisposition Syndrome
Status: Recruiting | Type: Observational
Sponsor: Mohamed Abdel-Rahman (Other)
Responsible Party: Sponsor-Investigator, Mohamed Abdel-Rahman, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2014C0072
Record Dates: First submitted 2021-03-07; First posted 2021-03-11 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Uveal Melanoma; Cutaneous Melanoma; BAP1 Gene Mutation; Renal Cell Carcinoma; Mesothelioma; Hepatocellular Carcinoma; Cholangiocarcinoma; Meningioma Atypical
MeSH Terms: conditions — Uveal Melanoma; Melanoma; Carcinoma, Renal Cell; Mesothelioma; Carcinoma, Hepatocellular; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with personal and/or family history suggestive of hereditary BAP1: Personal history of one cancer reported in BAP1 cancer predisposition syndrome and family history of at least two 1st or 2nd degree relatives with cancer reported in hereditary BAP1 cancer predisposition syndrome such as UM, CM, mesothelioma, RCC, cholangiocarcinoma, hepatocellular carcinoma and meningioma
- Pathogenic, likely pathogenic variants in BAP1 and variants of uncertain significance: Affected and unaffected individuals with pathogenic or likely pathogenic variant in BAP1 and their family members
  Patients with personal family history of any of the BAP1 associated cancer and a variant of uncertain significance of BAP1

SUMMARY:
This research will have a significant impact on the overall management of those cancer patients and their family members who are at risk for hereditary cancer due to germline inactivation of BAP1. Our study will ultimately facilitate the development of novel screening, prevention and treatment strategies for these individuals with the syndrome. Because the vast majority of UM develop in pre-existing nevi, characterization of individuals at high risk for development of UM will allow closer screening and earlier intervention which would improve the treatment outcome not only for retaining vision but also for overall survival. Similarly in patients with germline BAP1 mutation CM develops in premalignant atypical melanocytic lesions and careful follow up of these patients will improve the outcome of their disease. In addition this study could have impact on the management of patients with personal and/or family history of several other cancers reported in patients with germline BAP1 mutation such as mesothelioma, renal cell carcinoma, cholangiocarcinoma, hepatocellular carcinoma, meningioma and basal cell carcinoma.

DETAILED DESCRIPTION:
BAP1 (BRCA1-associated protein-1), is a deubiquitinating enzyme with a ubiquitin carboxy-terminal hydrolase function that has been suggested to be a tumor suppressor gene with a role in cell proliferation and growth inhibition. Recently germline mutations in BAP1 have been identified by our group and others in families with hereditary cancers. However, the clinical spectrum of cancers in patients with germline BAP1 is still not clear. The association of germline BAP1 mutations with increased risks for uveal melanoma (UM), mesothelioma, cutaneous melanoma (CM), renal cell carcinoma (RCC) and BAP1-inactivated melanocytic tumors is fairly well established. However, several other cancers have been reported in these patients and their family members including cholangiocarcinoma, hepatocellular carcinoma, meningioma, basal cell carcinoma and other internal malignancies. Identification of the clinical phenotype of BAP1-TPDS is important for proper counseling and management of patients.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet any of the following criteria:

1. Personal history of one cancer reported in BAP1 cancer predisposition syndrome and family history of at least two 1st or 2nd degree relatives with cancer reported in hereditary BAP1 cancer predisposition syndrome such as UM, CM, mesothelioma, RCC, cholangiocarcinoma, meningioma and hepatocellular carcinoma.
2. Any patient with personal history of at least 2 cancers reported in hereditary BAP1 cancer predisposition syndrome.
3. Any subject (affected or unaffected) with a documented BAP1 pathogenic/ likely pathogenic variant.
4. Any patient with a cancer reported in BAP1 and a germline variant of uncertain significance.
5. At risk relatives of a patient with documented BAP1 mutation.

Exclusion Criteria:

* Study material including consent forms are currently only available in English so non-English speaking subjects are excluding

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Providers at OSU will identify eligible participants through clinical practice. Providers at other institutions who become aware of our research through presentations at conferences, publications, etc. may identify one of their patients as eligible or potentially eligible for the study and introduce the study to their patient.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-03-03 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of germline BAP1 variants in the unselected general population of cancer patients | 5 years
  Frequency of germline BAP1 pathogenic/likely pathogenic variants in different cancers
Clinical phenotypes (this includes premalignant lesions, tumor type and age of onset) in at risk blood-line family members of the patients | 5 years
  Questionnaire and chart review of the clinical phenotype

SECONDARY OUTCOMES:
Questionnaire to assess environmental risk factors modifying cancer risk in patients | 10 years
  Measurement used: questionnaire for various environmental risk factors
Genotyping to assess genetic risk factors modifying risk of cancer | 10 years
  Genotyping for genetic variants that could modify the risk of cancer in subjects.
Disease outcome (response to treatment, prognosis including prognostic markers) | 10 years
  Chart review of disease outcome
Tumor pathology and genomics (including tumor grade, stage, somatic genomic alterations) | 10 years
  Review of pathology and study of genomics alterations in tumors
Assessment of disease penetrance and life time risk estimate | 10 years
  Statistical assessment of disease penetrance and life time risk estimates of various cancers

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Abdel-Rahman, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No